CLINICAL TRIAL: NCT02258594
Title: Transforming the Acute Care Environment: BWH PROSPECT Framework
Brief Title: Promoting Respect and Ongoing Safety Through Patient-centeredness, Engagement, Communication and Technology
Acronym: PROSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Principal Investigator, David W. Bates, MD, MSc, Chief, Division of General Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013P001966
Record Dates: First submitted 2014-10-01; First posted 2014-10-07 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Medical Intensive Care Unit (MICU) Patients; Oncology Unit Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline - Usual Care (No Intervention): Usual Care on two Medical Intensive Care Units units
  Usual Care on four Oncology units
- Post-Implementation - Intervention Units (Experimental): PROSPECT Intervention (Web-Based Patient Centered Toolkit (PCTK) + The Patient-SatisfActive® Model) on two MICU units
  PROSPECT Intervention (Web-Based Patient Centered Toolkit (PCTK) + The Patient-SatisfActive® Model) on two Oncology units
  Interventions: Other: Web-Based Patient Centered Toolkit (PCTK); Behavioral: The Patient-SatisfActive® Model
- Post-Implementation - Usual Care (No Intervention): Usual Care on two Oncology Units

INTERVENTIONS:
Other: Web-Based Patient Centered Toolkit (PCTK) — The PCTK provides patients/care partners tailored health information regarding conditions, test results, and medications presented at a consumer health literacy level, and the ability to communicate with care team members via "patient-facing" tools accessible from bedside tablet computers. The PCTK allows patients to post questions to their care team members via a patient-centered microblog. The microblog facilitates development of a collaborative patient plan of care. The "provider-facing" PCTK includes tools that engage care team members in 1) completing a safety checklist and viewing a safety dashboard; 2) viewing patient-inputted information (goals, preferences, concerns) regarding the plan of care; 3) identifying clinical problems, care team goals, and patient schedules for education and multidisciplinary communication; 4) messaging patients on the "patient thread"; and 5) discussing patient's plan of care with other providers via the "provider thread".
  Arms: Post-Implementation - Intervention Units
Behavioral: The Patient-SatisfActive® Model — The Patient-SatisfActive Model is a structured, pro-active, patient-centered care model that aims at improving patient satisfaction by enhancing the degree to which patients' needs, concerns and expectations are met and by preserving dignity and respect. The model comprises steps that enhance interpersonal communication between clinicians and patients, incorporates clinicians' efforts to ascertain, address and document patients' needs, concerns, expectations and perceptions throughout hospitalization, and includes elements that empower and engage patients in their care.
  Arms: Post-Implementation - Intervention Units

SUMMARY:
The purpose of this project is to refine, implement, and evaluate a multi-component intervention that achieves sustainable and meaningful impact on healthcare quality, safety, and costs while ensuring dignity and respect for adult oncology and intensive care patients and their care partners. The PROSPECT (Promoting Respect and Ongoing Safety through Patient-centeredness, Engagement, Communication, and Technology) framework will achieve this by enhancing the patient-provider relationship and introducing patient-centered approaches to multi-disciplinary communication and patient education. The PROSPECT framework is based upon a validated structured, team-work training model and novel web-based technology. The overarching goals of this project are to achieve the following:

1. Optimize the overall experience of patients (including their family/care partners) by promoting dignity/respect, encouraging engagement, improving care plan concordance, and enhancing satisfaction.
2. Minimize preventable harms in two environments: intensive care and acute care oncology units.
3. Reduce unnecessary healthcare resource utilization and associated costs.

DETAILED DESCRIPTION:
This overarching project aims are to refine, implement, and evaluate a multi-faceted intervention composed of the Patient-SatisfActive® model, developed by Drs. Ronen Rozenblum and David Bates at Brigham and Women's Hospital, and a web-based Patient-Centered Toolkit (PCTK), developed by Drs. Dykes and Dalal, on quality, safety, and cost outcomes in the intensive care and oncology units at Brigham and Women's Hospital. The specific aims of the project are as follows:

* Aim 1: To refine and implement the Patient-SatisfActive® model to promote respect, dignity, and satisfaction of patients, care partners and staff on intensive care and oncology units.
* Aim 2: To refine and implement a web-based, Patient-Centered Toolkit (PCTK), comprised of an electronic bedside communication center (eBCC) and a patient-centered microblog, to promote tailored patient and care-partner education, communication, collaboration, and engagement.
* Aim 3: To evaluate the relative impact of this intervention compared to usual care on patient reported outcome measures, adverse events (harms), post-discharge healthcare utilization, concordance in understanding the care plan, and satisfaction among care team members (patients/care partners, profession providers).
* Aim 4: To identify the barriers and facilitators of implementing this intervention to support dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Any patient admitted or transferred to designated care units
* Admitted or transferred to a MICU or Oncology service
* On the designated unit for at least 24 hours

Exclusion Criteria:

* Age < 18
* Any patient admitted or transferred to designated care unit but NOT on a MICU or Oncology service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4368 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Preventable Harms (Adverse Events) in the Acute Care Setting | Enrolled patients will be followed for the duration of hospital stay, typically ranging from 5 to 30 days.
  Preventable adverse events in the acute care setting include medication errors, patient falls, veno-thromboembolism, hospital acquired infection, central line related bloodstream infection, ventilator associated pneumonia, catheter associated urinary tract infection, newly acquired physical harm/injury. We will measure the rate of adverse events acquired from the time of admission to study units through hospital discharge. Using an adaptation of the Institute for Healthcare Improvement (IHI) Global Trigger Tool, we will randomly sample charts of enrolled patients from intervention and control units during the pre-intervention and post-intervention periods to identify adverse events. The length of hospital stay for patients admitted to medical intensive care and oncology units at our institution is variable, typically ranging from 5 to 30 days.

SECONDARY OUTCOMES:
Patient Experience & Satisfaction & Engagement | At time of transfer/discharger from study unit and up to 45-days post-hospitalization
  Randomly selected patients transferred from the MICU units will receive FS-ICU survey, semi-structured interviews, and 45-day post-hospitalization phone survey
  Randomly selected patients discharged from Oncology units will receive semi-structured interviews and 45-day post-hospitalization phone survey. Data from national patient satisfaction survey, HCAHPS, will be collected and analyzed.
Healthcare Resource Utilization | From time of hospital admission through 30-days post-discharge
  Inpatient healthcare utilization measures: Total cost of hospitalization and hospital length of stay (total, ICU, and non-ICU) from administrative data for each enrolled patient.
  Post-discharge healthcare utilization measures: Rate of unscheduled utilization of health care resources (ambulatory/urgent care visits, emergency room visits, hospital readmissions) during the 30-day post-discharge period using the combination of administrative data and patient reports during their 30-day interview.
Care Plan Concordance | Approximately 48-72 hours after admission to study unit
  Structured interviews (9-question survey) with patient/care partners, a member of the inpatient medical team (attending, resident, or intern), inpatient nurses, and one additional care team member (e.g., PCP, ambulatory specialists) will be conducted after admission to MICU or Oncology units. Concordance for each item of survey will be rated on a 3-point scale (0, 1, 2) for each dyad. The scores of all dyads will be summed as a global concordance score for each patient.
Perceptions of Communication/Collaboration | Once during baseline (pre-intervention) and post-intervention periods, approximately 12 months
  Overall perception of collaboration and satisfaction with communication among the various members of the care team will be measured on a 5-point Likert scale via surveys administered during the baseline and intervention periods. Scores will be dichotomized.
Patient Safety Climate | Once during baseline (pre-intervention) and post-intervention periods, approximately 12 months
  The AHRQ Patient Safety Culture (PSC) survey will be used to control for differences across units and facilities that may impact incidence of adverse events (communication, leadership, teamwork, frequency of reporting, perceived patient safety score).
Dignity and Respect | At time of transfer/discharger from study unit and up to 45-days post-hospitalization
  Randomly selected patients transferred from the MICU will receive the FS-ICU survey, which contains several questions related to dignity and respect. Randomly selected patients will also receive semi-structured interviews to enhance understanding of dignity and respect.
  Randomly selected patients discharged from Oncology units will receive semi-structured interviews regarding perceptions of dignity and respect and a 45-day post-hospitalization phone survey. Relevant data from national patient satisfaction survey, HCAHPS, will be collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: David W Bates, MD, MSc, Principal Investigator — Brigham and Women's Hospital; Patricia Dykes, RN, DNSc, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dalal AK, Dykes P, Samal L, McNally K, Mlaver E, Yoon CS, Lipsitz SR, Bates DW. Potential of an Electronic Health Record-Integrated Patient Portal for Improving Care Plan Concordance during Acute Care. Appl Clin Inform. 2019 May;10(3):358-366. doi: 10.1055/s-0039-1688831. Epub 2019 May 29. PMID 31141830
- [Derived] Gazarian PK, Morrison CRC, Lehmann LS, Tamir O, Bates DW, Rozenblum R. Patients' and Care Partners' Perspectives on Dignity and Respect During Acute Care Hospitalization. J Patient Saf. 2021 Aug 1;17(5):392-397. doi: 10.1097/PTS.0000000000000353. PMID 28230575